CLINICAL TRIAL: NCT07287267
Title: Exploring the Relationship Between Range of Motion in Knee Rehabilitation Exercises and Pain in Patellofemoral Pain Syndrome
Status: Recruiting | Type: Observational
Sponsor: Ted Gunhamn (Other)
Responsible Party: Sponsor-Investigator, Ted Gunhamn, PhD Candidate, Linnaeus University
Organization: Linnaeus University (Other)
Other Study IDs: 2024-01422-01
Record Dates: First submitted 2025-09-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Patello Femoral Syndrome
Keywords: Patellofemoral pain syndrome; Range of motion; patellofemoral pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patellofemoral Pain Syndrome: Patients diagnosed with patellofemoral pain syndrome by health care provider.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise with progressively increased range of motion.

SUMMARY:
This study aims to investigate the relationship between knee joint range of motion and pain in patients with patellofemoral pain syndrome (PFPS). In a cross-sectional observational design, PFPS patients will perform trials involving progressively increased knee joint range of motion in three closed-chain exercises: squat, single-leg squat, and split squat. During each trial, participants will report pain levels on a 0-10 Visual Analog Scale (VAS) until either (1) achieving full depth in the respective exercise or (2) reaching a pain level of >5 on the VAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PFP in only one knee by a licensed healthcare professional.
* Aged 15-35 years.
* A physical activity level of 3/10 or higher on the Tegner Activity Scale before the injury.

Exclusion Criteria:

* Any prior injury or condition with residual symptoms that may affect the results.
* Current injury or condition affecting the performance of the test.
* Resting pain greater than 0-1/10 on the Numeric Pain Rating Scale (NRS) and pain greater than 1-2/10 during light daily activities such as walking, sitting, standing, or climbing stairs.

Ages: 15 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: This project will include patients diagnosed with PFP (ICD-10: M22.2).
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS) | Day 1 (Cross sectional single session. Outcomes will be collected during one single session for each participant.)
  Pain measured 0-10 visual analog scale (VAS) reported during each trial of progressively increased range of motion during a single session.
Range of motion | Day 1 (Cross sectional single session. Outcomes will be collected during one single session for each participant.)
  Degrees of knee flexion measured during each trial in one single session.

SECONDARY OUTCOMES:
Force | Day 1 (Cross sectional single session. Outcomes will be collected during one single session for each participant.)
  Force (N) (peak value) reported during the different trials in one session. Measured by force plates.
Tegner Activity Scale (TAS) | Baseline (Administered at the beginning of the study)
  The Tegner Activity Scale (TAS) will be used to assess the physical activity levels of the participants. Scale from 1-10 where 10 is highest possible physical activity and 1 is sedentary.

CONTACTS AND LOCATIONS:
Locations (1):
- Linnaues University, Kalmar, Sweden